CLINICAL TRIAL: NCT07157917
Title: Translation and Application of the Chinese Thirst Safety Management Protocol: A Randomized Controlled Trial With Cultural Equivalence Validation Between Taiwan and Brazil
Brief Title: Thirst Translation and RCT
Acronym: SEDE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University (Other)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, Han-Yi Tsai, Taipei Medical University, School of Nursing, College of Nursing, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202508163RIN
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Thirst in Intensive Care Unit (ICU) Practice
Keywords: Thirst

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SEDE Group (Experimental): Intervene with a thirst management protocol
  Interventions: Other: Protocol based
- Usual care control (Placebo Comparator): Room temperature water if needed
  Interventions: Other: Control

INTERVENTIONS:
Other: Protocol based — Apply a thirst safety management protocol
  Arms: SEDE Group
Other: Control — Room air water
  Arms: Usual care control

SUMMARY:
To translate the SEDE-E (Extubated) and SEDE-T(tracheotomized) protocols-Chinese version and validate it with an RCT trial

ELIGIBILITY:
Inclusion Criteria:

1. Patients whose physicians have issued orders for removal of the endotracheal tube or who have undergone tracheotomy,
2. patients with clear consciousness
3. patients who can communicate in Chinese as their native language

Exclusion Criteria:

1. patients with water restriction
2. patients who have undergone thirst quenching intervention measurements in the recovery room.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Thirst intensity visual analogue scales | 0, 15, 60 minutes
  This is a 0~10 point Likert scale, with 0 indicates no thirsty, and 10 indicates the most severe thirsty.

IPD SHARING:
Plan to Share IPD: No
Patient private consideration